CLINICAL TRIAL: NCT05724186
Title: Clinical Evaluation of a Myopia Control Lens in Slowing Myopia Progression - Contiguous Spherical Lenslet
Brief Title: Clinical Evaluation of a Myopia Control Lens in Slowing Myopia Progression (CSL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WS10314
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Myopia
Keywords: refractive error; eye disease
MeSH Terms: conditions — Myopia; Refractive Errors; Eye Diseases

STUDY DESIGN:
Intervention Model Description: This is a mono-centre, prospective, one-arm, unmasked clinical trial, which consists of 6 visits, across 12 months. The objective of this clinical trial is to compare the test myopia control spectacle lens to the single vision control spectacle lens from the previous clinical trial, otherwise termed as historical control group.
  After obtaining informed consent and assent, a comprehensive eye examination will be conducted during the screening visit on all 40 myopic children between the age of 8 to 13 years old. Eligible children will return in a separate visit (baseline visit) to collect the study spectacles and the assessment of study spectacles, biometry and instructions to use study spectacles are established in the same visit. A follow up visit will be conducted in 3, 6 and 12 months time, where 12 months is the end of study. All of the eye examinations and assessments are non-contact and non-invasive to the eyes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test myopia control lenses (CSL) (Experimental): A pair of myopia control spectacle lenses (test lenses) will be given to subjects to wear for 12 months
  Interventions: Device: Test myopia control lenses (CSL)

INTERVENTIONS:
Device: Test myopia control lenses (CSL) — A pair of myopia control spectacle lenses (test lenses) will be given to subjects to wear for 12 months

SUMMARY:
This is a mono-centre, prospective, one-arm, unmask clinical trial to evaluate the effectiveness of test lens in slowing myopia progression with respect to axial length elongation compared to a single vision spectacle lens from the historical control group of another clinical trial NCT05331378. A total of 40 children will be recruited.

DETAILED DESCRIPTION:
As myopia is a growing worldwide problem, it is important to better understand the range of possible treatments to slow the progression of myopia. Spectacle lenses with aspherical lenslets were shown to be effective in reducing myopia progression and axial length elongation in children in the previous clinical trial (Bao et al. 2022). A dose-dependent effect was demonstrated, with higher lenslet asphericity having greater myopia control efficacy.

This open clinical trial will test the safety and effectiveness of a test lens designed to modify the area and amount of myopic defocus on the retina without compromising vision. The study population includes children in Singapore aged 8 to 13 years (40 subjects) at the time of commencing treatment. Axial length and spherical equivalent refraction will be the primary measure for myopia progression. Visual acuities will also be compared between test lenses and control lenses of the historical control group to determine the quality of vision using test lenses

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subject and guardian, fluent English spoken, willing to follow protocol and able to read, comprehend and sign the informed consent & assent form.
* 8 to 13 years old at time of informed consent and assent.
* Spherical equivalent refractive error (SER) by manifest refraction between -0.75 and -4.75 D in each eye.
* Astigmatism, if present, of not more than 1.50 D.
* Difference in SER between the two eyes (Anisometropia) by manifest refraction not more than 1.00 D.
* Best corrected visual acuity in each eye equal to or better than +0.10 logMAR (≥ 20/25 as Snellen)
* Be in good general health based on his/her and parent's/guardian's knowledge. Absence of ocular disease with full ophthalmic examination. Without any ocular or systemic condition known to affect refractive status.
* Absence of strabismus by cover test at near or distance wearing correction.
* Absence of amblyopia
* Without ocular or systemic medications which, in the investigator's opinion, may significantly affect pupil size, accommodation or refractive state.

Exclusion Criteria:

* Vulnerability of subject
* History of myopia control intervention
* Participation in any clinical study within 30 days of the Baseline visit.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Axial Length | 12 months
  Change in ocular axial length (mm) measured using Lenstar Optical Biometer.

SECONDARY OUTCOMES:
Spherical Equivalent Refraction | 6 months and 12 months
  Change in spherical equivalent refraction (Dioptres) through manifest subjective refraction.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tan, Principal Investigator — Essilor R&D Centre Singapore
Locations (1):
- Essilor R&D Centre Singapore, Singapore, Singapore

REFERENCES:
- [Background] Bao J, Yang A, Huang Y, Li X, Pan Y, Ding C, Lim EW, Zheng J, Spiegel DP, Drobe B, Lu F, Chen H. One-year myopia control efficacy of spectacle lenses with aspherical lenslets. Br J Ophthalmol. 2022 Aug;106(8):1171-1176. doi: 10.1136/bjophthalmol-2020-318367. Epub 2021 Apr 2. PMID 33811039